CLINICAL TRIAL: NCT00387725
Title: A Randomized, Observer-blinded, Parallel-group, Active-control, Phase ½ Trial Of The Safety, Immunogenicity, And Tolerability Of 20 Mg, 60 Mg, And 200 Mg Of Meningococcal Group B Rlp2086 Vaccine In Healthy Children And Adolescents Aged 8 To 14 Years
Brief Title: Study Evaluating Safety & Immunogenicity of rLP2086 Vaccine in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6108A1-501; B1971006 (Other: Alias Study Number)
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Adolescent; Meningococcal; Safety
MeSH Terms: interventions — factor H-binding protein, Neisseria meningitidis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): 20ug Experimental
  Interventions: Biological: rLP2086
- Group 2 (Experimental): 60ug Experimental
  Interventions: Biological: rLP2086
- Group 3 (Experimental): 200ug Experimental
  Interventions: Biological: rLP2086
- Group 4 (Active Comparator): Active comparator
  Interventions: Biological: rLP2086

INTERVENTIONS:
Biological: rLP2086 — Vaccine administered at 0, 1, and 6 months
  Arms: Group 4
Biological: rLP2086 — Vaccine administered at 0, 1, and 6 months
  Arms: Group 3
Biological: rLP2086 — Vaccine administered at 0, 1, and 6 months
  Arms: Group 2
Biological: rLP2086 — Vaccine administered at 0, 1, and 6 months
  Arms: Group A

SUMMARY:
Study to evaluate the safety of an investigational meningitis vaccine and the immune response to it in adolescents

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

* Aged 8 to 14 years at the time of enrollment.
* Healthy male or female subjects
* Negative urine pregnancy test for female subjects

Exclusion Criteria:

Exclusion Criteria

* Prior vaccination with a meningococcal B vaccine
* Prior meningococcal disease

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Australia (9):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Herston, Queensland
  - Princess Margaret Hospital for Children, Subiaco, Western Australia
  - Sir Albert Sakzewski Virus Research Centre (SASVRC), Herston
  - Women's & Children's Hospital, North Adelaide
  - The Telethon Institute for Child Health Research, Subiaco
  - National Centre for Immunisation, Westmead
  - Department of Paediatrics and Child Health, Woden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6108A1-501&StudyName=Study%20Evaluating%20Safety%20%26%20Immunogenicity%20of%20rLP2086%20Vaccine%20in%20Adolescents

RESULTS

PARTICIPANT FLOW:
Groups:
- Twinrix; Initial Formulation rLP2086 20 mcg; Initial Formulation rLP2086 60 mcg; Initial Formulation rLP2086 200 mcg: Given on a 0, 1-, 6- month schedule
Period: Overall Study
Arm/Group | Twinrix | Initial Formulation rLP2086 20 mcg | Initial Formulation rLP2086 60 mcg | Initial Formulation rLP2086 200 mcg
Started | 21 | 16 | 45 | 45
Completed | 20 | 15 | 43 | 43
Not Completed | 1 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Parent/legal guardian request | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Twinrix | Initial Formulation rLP2086 20 mcg | Initial Formulation rLP2086 60 mcg | Initial Formulation rLP2086 200 mcg | Total
Number analyzed (Participants) | 21 | 16 | 45 | 45 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.19 (1.44) | 10.69 (0.95) | 10.31 (1.24) | 10.31 (1.29) | 10.34 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 22 | 28 | 69
  Male | 11 | 7 | 23 | 17 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion in rLP2086 Specific Serum Bactericidal Assay (SBA) Titer 1 Month After Dose 2
Time Frame: 1 month after Dose 2
Measure: Number; unit: percentage of participants
Arm/Group | Twinrix | Initial Formulation rLP2086 20 mcg | Initial Formulation rLP2086 60 mcg | Initial Formulation rLP2086 200 mcg
Number analyzed (Participants) | 21 | 16 | 45 | 45
percentage of participants
  PMB1745 (N=19, 15, 44, 42) | 0.0 [0.0 to 17.6] | 33.3 [11.8 to 61.6] | 63.6 [47.8 to 77.6] | 83.3 [68.6 to 93.0]
  PMB17 (N=18, 16, 44, 42) | 0.0 [0.0 to 18.5] | 18.8 [4.0 to 45.6] | 52.3 [36.7 to 67.5] | 61.9 [45.6 to 76.4]

2. Primary Outcome: Percentage of Participants With Seroconversion in rLP2086 Specific SBA Titer 1 Month After Dose 3
Time Frame: 1 month after Dose 3
Measure: Number; unit: percentage of participants
Arm/Group | Twinrix | Initial Formulation rLP2086 20 mcg | Initial Formulation rLP2086 60 mcg | Initial Formulation rLP2086 200 mcg
Number analyzed (Participants) | 21 | 16 | 45 | 45
percentage of participants
  PMB1745 (N=19, 16, 41, 43) | 0.0 [0.0 to 17.6] | 68.8 [41.3 to 89.0] | 70.7 [54.5 to 83.9] | 90.7 [77.9 to 97.4]
  PMB17 (N=18, 16, 41, 43) | 0.0 [0.0 to 18.5] | 87.5 [61.7 to 98.4] | 82.9 [67.9 to 92.8] | 95.3 [84.2 to 99.4]

3. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Time Frame: Dose 1 up to 1 month after Dose 3
Measure: Number; unit: percentage of participants
Arm/Group | Twinrix | Initial Formulation rLP2086 20 mcg | Initial Formulation rLP2086 60 mcg | Initial Formulation rLP2086 200 mcg
Number analyzed (Participants) | 21 | 16 | 45 | 45
percentage of participants | 90.5 | 93.8 | 93.3 | 97.8

ADVERSE EVENTS:
Time Frame: Dose 1 up to 1 month after Dose 3
Arm/Group | Twinrix | Initial Formulation rLP2086 20 mcg | Initial Formulation rLP2086 60 mcg | Initial Formulation rLP2086 200 mcg
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/16 | 3/45 | 3/45
Other Adverse Events (participants affected / at risk) | 19/21 | 15/16 | 42/45 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix (N=21) | Initial Formulation rLP2086 20 mcg (N=16) | Initial Formulation rLP2086 60 mcg (N=45) | Initial Formulation rLP2086 200 mcg (N=45)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix (N=21) | Initial Formulation rLP2086 20 mcg (N=16) | Initial Formulation rLP2086 60 mcg (N=45) | Initial Formulation rLP2086 200 mcg (N=45)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 5
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0
Eyelid disorder (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 8 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3 | 3
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site movement impairment (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 3 | 1
Vessel puncture site reaction (General disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 5
Enterobiasis (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 5 | 5
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0
Infected bites (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 6 | 4
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 2 | 3 | 3
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1 | 4 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 5 | 25 | 23
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Viraemia (Infections and infestations) | 1 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 5 | 6
Viral upper repiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 3
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 4
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 4
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 1
Vaccination Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Venomous sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lymph node Palpable (Investigations) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 4
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 3
Headache (Nervous system disorders) | 12 | 4 | 18 | 23
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 10 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.